CLINICAL TRIAL: NCT02132923
Title: Prospective Study in Japanese Children Hospitalized With Respiratory Syncytial Virus Related Lower Respiratory Tract Infections
Brief Title: A Study in Japanese Children Hospitalized With Respiratory Syncytial Virus Related Lower Respiratory Tract Infections
Status: Completed | Type: Observational
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Other Study IDs: CR103420; ObserveRSV0002 (Other: Janssen R&D Ireland)
Record Dates: First submitted 2014-05-06; First posted 2014-05-07 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Respiratory Syncytial Virus
Keywords: Respiratory syncytial virus; RSV; Lower respiratory tract infection; LRTI; Acute respiratory infection; Japanese children

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with respiratory syncytial virus (RSV) infection: The RSV infection is laboratory confirmed
  Interventions: Biological: No intervention

INTERVENTIONS:
Biological: No intervention — This is an observational study. The children hospitalized with lower respiratory tract infection (LRTI) with a laboratory confirmed RSV infection will be monitored for maximum 7 days or until hospital discharge.

SUMMARY:
The purpose of the study is to assess viral kinetics and clinical symptoms kinetics of Respiratory Syncytial Virus (RSV) in pediatric patients hospitalized with RSV confirmed lower respiratory tract infection (LRTI).

DETAILED DESCRIPTION:
This is an exploratory prospective study (a study in which the patients are identified and then followed forward in time for the outcome of the study). The study will consist of two phases: a screening phase (Day 1) and an assessment phase (Day 2 to Day 7). During screening phase, pediatric patients consecutively hospitalized with RSV-related infection will be enrolled in the study within 24 hours of admission if symptomatic for maximum 5 days before the hospital admission and if the informed consent form (ICF) was obtained. The diagnosis of RSV infection will follow using a standard of care (SOC) rapid point point of care (POC) detection method available in the hospital unit on nasal specimens .During the assessment phase the collection of nasal specimens will be done daily for a maximum of 6 days (Day 2 to Day 7 of hospitalization) or until patients will be discharged from hospital. Approximately 50 patients will be enrolled in this study. The total duration of the study for each patient will be approximately 7 days. The study duration will extend until the targeted number of 50 RSV hospitalized children have completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Legal representative has provided Ethics Committee approved written informed onsent prior to any study-related procedure(s) being performed and is willing to allow the participation of child to the study for 7 consecutive days or until hospital discharge (whatever comes first)
* Patient hospitalized with lower respiratory tract infection (LRTI) during respiratory syncytial virus (RSV) epidemics, within 24h of hospitalization. The diagnosis of LRTI will follow the standard medical procedure in the hospital unit
* Onset of acute respiratory symptoms was less than or equal to 5 days ago
* Patient is RSV positive based on a rapid point of care (POC) detection method. The diagnosis of RSV infection will follow the standard medical procedure in the hospital unit

Exclusion Criteria:

- Patient does not fulfill the inclusion criteria

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients hospitalized with a laboratory confirmed Respiratory Syncytial Virus (RSV) lower respiratory tract infection.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2013-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Respiratory Syncytial Viral Load (rate of viral clearance) | Day 1 (baseline) to Day 3
  RSV viral clearance, defined as the change in log viral load (VL) from Day 1 to Day 3, where the VL is measured in nasal specimens with quantitative reverse transcript poly cycle reaction (qRT-PCR).

SECONDARY OUTCOMES:
Change From Baseline in Clinical Symptoms Score (CSS) | Day 1 (baseline) to Day 3
  The severity of the RSV disease will be assessed using CSS. CSS will be computed based on clinical parameters (O2 saturation, heart rate, respiratory rate) and lung auscultation examination. CSS score ranges from 0 (best) to 15 (worst). Higher scores indicate worsening.
Change From Baseline in Medical Support Score (MSS) | Day 1 (baseline) to Day 3
  The severity of the RSV disease will be assessed using MSS. MSS will take into account the use of supplementary oxygen, the request for mechanical ventilation, intensive care unit admission and the length of hospitalization. The MSS score ranges from 0 (best) to 5 (worst). Higher scores indicate worsening.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (1):
- Tokyo, Japan